CLINICAL TRIAL: NCT02819349
Title: Texting for Relapse Prevention Among People Diagnosed With Schizophrenia or SAD
Brief Title: Texting for Relapse Prevention
Acronym: T4RP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Innovative Public Health Research (Other)
Collaborators: Johns Hopkins University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R34MH108781 (NIH); 1R34MH108781 (NIH)
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Relapse Prevention; People with Schizophrenia; Text-Messaging; Assertive Community Treatment (ACT)
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Secondary Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Texting for Relapse Prevention (T4RP) (Experimental): T4RP is a relapse prevention mHealth program text messaging to people who have schizophrenia/SAD. The intervention will include an online interface for clinicians and an automated text messaging program for patients. Firstly, patients and providers will meet in an intake session, to identify the patient's personal early warning signs from a pre-identified list. Using the online interface, providers will enter additional warning signs or personalize the wording of the messages as requested by the patient. The patient also will determine the threshold at which the provider will be alerted about a possible relapse and whether additional contact people should be alerted.
  Interventions: Behavioral: Texting for Relapse Prevention (T4RP)
- Treatment-As-Usual Control (No Intervention): The control group will be a treatment as usual comparison group. For the majority of individuals with schizophrenia/SAD in care at JHCPP, this involves meeting with their therapist every 2 to 4 weeks and meeting with their psychiatrist at least once every 90 days or more frequently as clinically indicated. All routine appointments are scheduled, but individuals can walk in or call if they do not feel well between sessions.

INTERVENTIONS:
Behavioral: Texting for Relapse Prevention (T4RP) — T4RP is a relapse prevention mHealth program text messaging to people who have schizophrenia/SAD. Content is guided by components of the Assertive Community Treatment (ACT) and focuses on facilitating improved patient-provider communication, promoting medication adherence, helping people self-monitor their early warning signs, and promoting self-management of symptoms.
  Arms: Texting for Relapse Prevention (T4RP)

SUMMARY:
The purpose of this study is to examine whether Texting for Relapse Prevention (T4RP), a text messaging-based early warming for relapse prevention in people who have schizophrenia/SAD, is associated with fewer relapse symptoms compared to a treatment-as-usual control group.

DETAILED DESCRIPTION:
Schizophrenia is among the 20 most debilitating illnesses worldwide, responsible for 1% of the global burden of disease. Schizoaffective disorder (SAD) affects an additional 0.2% to 1.1% of adults. As many as four out of five people who have schizophrenia or SAD relapse within 5 years of recovery from their initial episode. Interventions aimed at early intervention to prevent relapse would impact public health.

The Texting for Relapse Prevention (T4RP) is an innovative service delivery program delivered via text messaging designed for people who have schizophrenia/SAD. The intervention will be tested in a randomized controlled trial against a treatment-as-usual control group which, for most, involved meeting with their therapist every 2 to 4 weeks and meeting with their psychiatrist at least once every 90 days or more frequently as clinically indicated. A total of 40 people with schizophrenia and 5-15 provider participants (depending on the patient distribution across the providers) in the pilot RTC. The study is being conducted by researchers at the Center for Innovative Public Health Research and Johns Hopkins Community Psychiatry Program (JHCPP).

The investigators posit that T4RP will reduce psychiatric morbidity and institutionalization rates and promote recovery by facilitating improved patient-provider communication, promoting medication adherence, helping people self-monitor their early warning signs, and promoting self-management of symptoms.

If T4RP is effective, this cost-effective and easily scalable intervention will make a significant public health impact and reduction in relapse-related costs for people with schizophrenia/SAD.

ELIGIBILITY:
Inclusion Criteria:

* be English-speaking;
* have a chart diagnosis of schizophrenia or SAD
* be able to provide consent (i.e., pass the Capacity to Consent screen)
* own a cell phone and report using the text messaging function
* be currently at their personal baseline with regard to symptoms and functioning as assessed by their provider (i.e., not in relapse and compliant with treatment)
* be actively under the care of a mental health provider enrolled in the program
* agree to continue attending the clinic for the duration of the study
* plan to keep the same cell phone number for the duration of the study
* have at least one of their providers consent to take part in the study

Exclusion Criteria:

* have at least one of their providers consent to take part in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2019-04-09 (Actual)

PRIMARY OUTCOMES:
The Positive and Negative Syndrome Scale (PANSS) | 6-months post-study enrollment
  It has three subscales that measure: positive symptoms of schizophrenia, negative symptoms of schizophrenia, and general psychopathology.
Montgomery-Asberg Depression Scale (MADRS) | 6-months post-study enrollment
  It is a clinician-administered 10-item scale developed to measure changes in depressive symptom during treatment.
Young Mania Rating Scale (YMRS) | 6-months post-study enrollment
  It is is an 11-item clinician administered scale that assesses the presence and severity of manic symptoms.
Institutionalization | 6-months post-study enrollment
  The number of hospitalizations or ER crisis visits during the study period
Recovery Assessment Scale | 6-months post-study enrollment
  It is a 41-item self-report scale with 5 subscales that measure an individual's experience of recovery

SECONDARY OUTCOMES:
Brief Adherence Rating Scale | 6-months post-intervention
  It is a clinician-administered, 4-item scale that has three questions and an overall visual analog scale. It was designed for use in community settings with individuals who have schizophrenia or schizoaffective disorder and has been validated against electronically-monitored adherence.
Boston University Empowerment Scale | 6-months post-intervention
  It is a 28-item self-report scale that measures empowerment among those using mental health services.
Brief Cognitive Assessment | 6-months post-intervention
  It is a clinician administered test that consists of 3 standard tests: Verbal Fluency, Hopkins Verbal Learning Test and Trails A and B and has been shown to be related to measures of functional outcome in patients with schizophrenia.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Ybarra, PhD, Principal Investigator — Center for Innovative Public Health Research (CiPHR); Bernadette Cullen, PhD, Principal Investigator — Johns Hopkins Community Psychiatry Program (JHCPP)
Locations (1):
- Johns Hopkins Community Psychiatry Program (JHCPP), Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ybarra ML, Rodriguez K, Madison H, Mojtabai R, Cullen BA. Developing Texting for Relapse Prevention: A Scalable mHealth Program for People With Schizophrenia and Schizoaffective Disorder. J Nerv Ment Dis. 2019 Oct;207(10):854-862. doi: 10.1097/NMD.0000000000001037. PMID 31503175

DOCUMENTS (1):
  • Informed Consent Form (2017-12-04): https://cdn.clinicaltrials.gov/large-docs/49/NCT02819349/ICF_000.pdf